CLINICAL TRIAL: NCT02888028
Title: Quality of Life and Device Acceptance in Patients With Implantable Cardioverter-defibrillators Undergoing Remote ICD Follow-up
Brief Title: Quality of Life and Device Acceptance in Patients With ICD Undergoing Remote ICD FU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LMU Klinikum (Other)
Collaborators: Klinikum Bielefeld (Other)
Responsible Party: Principal Investigator, Johannes Siebermair, MD, Johannes Siebermair, MD, LMU Klinikum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE MucM001-11
Record Dates: First submitted 2014-07-03; First posted 2016-09-02 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Anxiety; Depression
Keywords: Remote ICD follow-up; HRQoL; Health related Quality of Life; Depression; anxiety; device acceptance; telemedicine; telemonitoring
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ICD remote monitoring (Active Comparator): Active Comparator: ICD remote monitoring additionally to regular in-office visits/FU 1,3,6 and 12 months post implantation of an ICD or post ICD replacement
  Interventions: Procedure: ICD remote monitoring
- Control group (Other): Regular in-office visits/FU 1,3,6 and 12 months post implantation of an ICD or post ICD replacement w/o remote FU
  Interventions: Other: Control group

INTERVENTIONS:
Procedure: ICD remote monitoring — ICD remote monitoring additionally to regular in-office visits
  Arms: ICD remote monitoring
Other: Control group — Regular in-office visits/FU 1,3,6 and 12 months post implantation of an ICD or post ICD replacement w/o remote FU
  Arms: Control group

SUMMARY:
This study investigates whether an additional remote follow-up of patients with implantable cardioverter-defibrillators (ICDs) has beneficial effects on Quality of life (QoL), levels of anxiety and depression and device acceptance. Patients are randomized to either conventional in-office FU only or additional remote surveillance, follow-up duration is 12 months. The influence of other variables (age, sex,..) is evaluated regarding their influence on study endpoints.

DETAILED DESCRIPTION:
The rising number of implantable cardiac devices leads to an increasing amount of device-related workload, e.g. regular in-office follow-ups (FU). New means of ICD FU strategies are necessary to handle the increasing burden. ICD remote monitoring promises a time- and cost efficient alternative to conventional in-office FU strategies. Many studies have already shown benefits on FU burden reduction, on saving of costs and time, and recently on total mortality. The impact of remote ICD FU on Quality of life, anxiety and depression levels and device acceptance is still under discussion. The aim of this trial is to investigate the influence of additional remote ICD surveillance on the primary endpoint health related quality of life (HRQoL), further on levels of anxiety and depression and on device acceptance.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to participate
* Patients with new-implantation of an ICD or device replacement due to battery depletion between May 2011 and April 2013
* Sufficient knowledge of the German language
* Expectancy of life >1 years at good clinical status
* Written informed consent

Exclusion Criteria:

* Age <18 years
* Subjects not able to give written informed consent
* Subjects without sufficient German language skills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2011-05; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Influence of ICD remote monitoring on Quality of Life, measured by the EQ5D questionnaire | 12 months

SECONDARY OUTCOMES:
Influence of ICD remote monitoring on levels of anxiety and depression, measured by the HADS questionnaire (Hospital Anxiety and Depression scale) | 12 months
Influence of ICD remote monitoring on device acceptance, measured by the Florida Patient acceptance scale (FPAS) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Siebermair, MD, Principal Investigator — Munich University Clinic, Campus Grosshadern, Munich, Germany; Florian Leppert, MSc, Principal Investigator — Bielefeld University, School of public health Bielefeld, Germany; Stefan Kääb, MD, Principal Investigator — Munich University Clinic, Campus Grosshadern, Munich, Germany; Wolfgang Greiner, MD, Principal Investigator — Bielefeld University, School of public health, Bielefeld, Germany
Locations (2):
- Germany (2):
  - Bielefeld University, School of public health, Bielefeld
  - Munich University Clinic, Campus Grosshadern, Munich

IPD SHARING:
Plan to Share IPD: No